CLINICAL TRIAL: NCT00173745
Title: Treatment of Drooling With Type A Botulinum Toxin A in Children With Cerebral Palsy
Brief Title: Treatment of Drooling With Type A Botulinum Toxin in Children With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 9100012973; NSC93-2614-B-002-005
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-12-21 (Estimated); Status verified 2002-07

CONDITIONS: Cerebral Palsy; Drooling
Keywords: cerebral palsy; drooling; botulinum toxin
MeSH Terms: conditions — Cerebral Palsy; Sialorrhea | interventions — Botulinum Toxins, Type A

INTERVENTIONS:
Drug: botulinum toxin A injection

SUMMARY:
The purpose of this study is to evaluate the effectiveness of botulinum toxin injection to treat drooling in children with cerebral palsy, and to find the most appropriate dosage, duration of effect and side effects.

DETAILED DESCRIPTION:
Sialorrhea, or drooling, has been reported to be a significant problem in 10%to 37% of patients with cerebral palsy. Excessive drooling may cause skin maceration, increased the burden of caregiver, affect articulation of the patients, and increase the risk of aspiration and dehydration. Many options, including various therapies, medications, surgeries and radiation, have been proposed to treat drooling. Yet none of these is universally successful and many have potential complications. Nerve endings of the parasympathetic post-ganglionic neurons secret aceylcholine. Botulinum toxin should be able to inhibit salivary gland secretion by blocking the release of acetylcholine. Very limited case series had proved fair result of botulinum toxin injection to treat drooling. However, most of the subjects were adult patients with neurological disorders. The purpose of this study is to evaluate the effectiveness of botulinum toxin injection to treat drooling in children with cerebral palsy, and to find the most appropriate dosage, duration of effect and side effects.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of cerebral palsy
* severe drooling
* aged 6-21 yrs
* subjects (or their guardian) who are able to understand the requirements of the study and sign the informed consent form

Exclusion Criteria:

* age below 6 yrs or above 21 yrs
* known allergy or sensitivity to the study medication or its component
* diagnosis of myasthenia gravis, amyotrophic lateral sclerosis or any other disease that might interfere with neuromuscular function
* subjects who have prior surgery of the submandibular gland
* subjects who are receiving medication that affect drooling such as anticholinergic drug
* inability to give informed consent

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20
Dates: Start 2003-06; Study Completion 2005-09

PRIMARY OUTCOMES:
the effectiveness of botulinum toxin in treatment of drooling

SECONDARY OUTCOMES:
the most appropriated dosage of treatment
duration of effect
side effects

CONTACTS AND LOCATIONS:
Overall Officials: Jeng Yi Shieh, MD, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University hospital, Taipei, Taiwan